CLINICAL TRIAL: NCT01272271
Title: Postmarket Study of the Safety of Overnight Corneal Reshaping Lenses
Brief Title: Safety of Overnight Corneal Reshaping Lenses
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Bausch & Lomb Incorporated (Industry); CooperVision, Inc. (Industry)
Responsible Party: Mark A. Bullimore, Professor, The Ohio State University
Other Study IDs: 2007H0273
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Keratitis; Myopia
Keywords: Contact lens; Infection; Cornea
MeSH Terms: conditions — Keratitis; Myopia; Infections; Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children
- Adults

SUMMARY:
This retrospective chart review study compares the incidence of corneal inflammation due to infection in children vs. adult patients wearing overnight corneal reshaping lenses.

ELIGIBILITY:
Inclusion Criteria:

* Patients completing at least 3 months of wearing corneal reshaping lenses

Exclusion Criteria:

* Less than 3 months of wearing corneal reshaping lenses

Ages: 5 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Randomized sample of optometry and ophthalmology patients seen by 200 practitioners in various practice settings, stratified on manufacturer, practitioner volume.
Sampling Method: Probability Sample
Enrollment: 1317 (Actual)
Dates: Start 2008-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Microbial keratitis incidence | 1 year
  Incidence of microbial keratitis in children vs. adults with the use of two brands of corneal reshaping lenses.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Bullimore, PhD, Principal Investigator — Ohio State University